CLINICAL TRIAL: NCT01650571
Title: Evaluation of a 'Hand-Held' Fluorescence Digital Imaging Device for Real-Time Advanced Wound Care Monitoring (SMH/UHN)
Acronym: SMH/UHN
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Cancer Care Ontario (Other)
Responsible Party: Sponsor
Other Study IDs: 12-5024-A
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Surgical Wounds
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Currently, standard wound care practice is suboptimal at assessing wound remodeling and bacterial infection in real-time. An alternative and complimentary means of providing real-time imaging of connective tissue re-modeling and bacterial infection may greatly increase the early detection of infection thus leading to rapid therapeutic intervention. Our new device, PRODIGI(TM), images tissue and bacterial autofluorescence (without agents) and may provide this clinically-important capability.

In preliminary preclinical testing, the investigators have discovered that when wounds are illuminated by violet/blue light, endogenous collagen in the connective tissue matrix emit a characteristic green fluorescent signal, while most pathogenic bacterial species emit a unique red fluorescence signal due to the production of endogenous porphyrins. Therefore, with autofluorescence imaging, no exogenous contrast agents are needed during imaging, making this approach particularly appealing as a diagnostic imaging method for clinical use.

The investigators hypothesize that real-time imaging of tissue autofluorescence signals emanating from endogenous connective tissue (e.g. collagen) and pathogenic bacteria within complex wounds can be used to determine healing status (i.e., collagen re-modeling and wound closure), detect wound bacterial contamination and/or infection that is occult under standard clinical white light evaluation, and guide intervention and wound care.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. males and females
3. receiving care as in-patient at St. Michael's Hospital
4. presenting with abdominal wounds resulting from general surgery with known or unknown infection status.

Exclusion Criteria:

1. treatment with an investigational drug within 1 month before study enrolment
2. any contra-indication to routine wound care and/or monitoring
3. inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with wounds resulting from general abdominal surgery will be entered into this trial, based on statistical power-based calculations for sample size determined in collaboration with the UHN Biostatistics Group (assuming one wound per patient).
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
providing wound healing status in real time based on collagen fluorescence as an indicator of wound closure | Upon study completion

SECONDARY OUTCOMES:
detecting bacterial contamination and infection in wounds that is occult to conventional wound assessment methods (white light visualization and clinical signs and symptoms of wound infection) | Upon study completion
the ability of the device to provide real-time fluorescence image-guided targeting of swabbing for bacteriology testing | Upon study completion
utility of PRODIGI™ in guiding intervention | Upon study completion

CONTACTS AND LOCATIONS:
Overall Officials: Ralph S DaCosta, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada